CLINICAL TRIAL: NCT00065507
Title: Comparison of the Efficacy and Safety of Entecavir Versus Adefovir in Subjects Chronically Infected With Hepatitis B Virus and Evidence of Hepatic Decompensation
Brief Title: Comparison of Entecavir to Adefovir in Chronic Hepatitis B Virus (HBV) Patients With Hepatic Decompensation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI463-048
Record Dates: First submitted 2003-07-28; First posted 2003-07-29 (Estimated); Results first posted 2010-07-02 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Hepatitis B
Keywords: hepatic decompensation
MeSH Terms: conditions — Hepatitis B | interventions — entecavir; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: Entecavir (ETV)
- A2 (Active Comparator)
  Interventions: Drug: Adefovir (ADV)

INTERVENTIONS:
Drug: Entecavir (ETV) — Tablets, Oral, 1 mg once daily, 96 weeks from the time the last patient is randomized
  Other Names: Baraclude; BMS-200475
  Arms: A1
Drug: Adefovir (ADV) — Tablets, Oral, 10 mg, once daily, 96 weeks from the time the last patient is randomized
  Arms: A2

SUMMARY:
This is a phase IIIb comparative study of entecavir 1.0 mg once daily (QD) vs. adefovir 10 mg QD in patients who have chronic hepatitis B infection and hepatic decompensation. The patients are treated for 96 weeks after the last subject is randomized.

ELIGIBILITY:
Inclusion

* Child-Pugh (CP) score >= 7
* Hepatitis B virus (HBV) viremia

Exclusion

* Alanine aminotransferase (ALT) > 15 x upper limit of normal (ULN)
* Human immunodeficiency virus (HIV)/hepatitis C virus (HCV)/hepatitis D virus (HDV) coinfection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2003-08; Primary Completion 2008-10 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (55):
- United States (16):
  - Research And Education, Inc., San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - University Of Miami School Of Medicine, Miami, Florida
  - Pediatric Gasteroenterology, Atlanta, Georgia
  - Hawaii Medical Center East, Honolulu, Hawaii
  - Indiana University Med Center, Indianapolis, Indiana
  - The Cht Liver Research Center, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Health System Irb, Detroit, Michigan
  - Mount Sinai Medical Center, New York, New York
  - Columbia Presbyterian Medical Center (Cpmc), New York, New York
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Baylor University Medical Center, Dallas, Texas
  - Ut Southwestern Medical Center, Dallas, Texas
  - Mcguire Dvamc, Richmond, Virginia
- Brazil (4):
  - Local Institution, Porto Alegre - Rs, Rio Grande do Sul
  - Local Institution, Sao Paulo - Sp, São Paulo
  - Local institution, São Paulo, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (2):
  - Local Institution, Calgary, Alberta
  - Local Institution, Vancouver, British Columbia
- France (2):
  - Local Institution, Clichy
  - Local Institution, Strasbourg
- Greece (4):
  - Local institution, Athens
  - Local Institution, Athens
  - Local Instituition, Thessaloniki
  - Local Institution, Thessaloniki
- Local Institution, Tai Po, Hong Kong
- India (4):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Kolkata
  - Local Institution, Lucknow
  - Local Institution, New Delhi
- Local Institution, Jakarta, Indonesia
- Philippines (2):
  - Local Institution, Cebu
  - Local Institution, Manila
- Poland (4):
  - Local Institution, Bydgoszcz
  - Local Institution, Chorzów
  - Local Institution, Krakow
  - Local Institution, Lodz
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Smolensk
- Local Institution, Singapore, Singapore
- South Africa (2):
  - Local Institution, Observatory, Western Cape
  - Local Institution, Paarl, Western Cape
- Taiwan (5):
  - Local Institution, Changhua
  - Local Institution, Taichung
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
  - Local Institution, Tianan
- Thailand (2):
  - Local Institution, Bangkok
  - Local Institution, Hat Yai
- Turkey (Türkiye) (2):
  - Local Institution, Adana
  - Local Institution, Izmir
- Local Institution, London, Greater London, United Kingdom

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 431 participants were enrolled into the study. 236 were never randomized (213 no longer met study criteria; 6 withdrew consent; 3 died; 1 for administrative reasons by sponsor; 1 for adverse events; 1 lost to follow-up; 11 for other reasons).
Groups:
- Entecavir (ETV) 1.0 mg: Tablets, Oral, 1 mg once daily
- Adefovir (ADV) 10 mg: Tablets, Oral, 10 mg once daily
Period: Overall Study
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Started | 100 (101 participants were randomized; 1 never treated.) | 91 (94 participants were randomized; 3 never treated.)
Treated (As-Randomized Population) | 100 (As-randomized population was used in efficacy analyses, unless otherwise noted.) | 91 (As-randomized population was used in efficacy analyses, unless otherwise noted.)
Treated (As-Treated Population) | 102 (2 subjects randomized to ADV were treated with ETV for the entire dosing period and included in ETV.) | 89 (2 subjects randomized to ADV were treated with ETV for the entire dosing period and included in ETV.)
Treated, Wk 48 (As-Treated Population) | 102 (2 subjects randomized to ADV were treated with ETV for the entire dosing period and included in ETV.) | 89 (2 subjects randomized to ADV were treated with ETV for the entire dosing period and included in ETV.)
Treated, 24-Week Follow-Up Population | 25 | 28
Completed | 71 (Completed first 48 weeks of treatment) | 62 (Completed first 48 weeks of treatment)
Not Completed | 29 | 29
Not completed — Death | 16 | 17
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 0 | 6
Not completed — Poor/Non-compliance | 3 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Subject Withdrew Consent | 2 | 1
Not completed — Subject No Longer Meets Study Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg | Total
Number analyzed (Participants) | 100 | 91 | 191
Age Continuous [Mean (Standard Deviation); unit: years] | 51 (12) | 53 (11) | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 49
  Male | 78 | 64 | 142
Race/Ethnicity, Customized [Number; unit: participants] — Other category includes Asian Indian, South African "color," "mixed ancestry," and "mixed race"
  participants
    Asian | 55 | 49 | 104
    White | 35 | 28 | 63
    Other | 5 | 9 | 14
    Black/African American | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21
  Philippines | 4 | 5 | 9
  Taiwan | 11 | 11 | 22
  Hong Kong | 5 | 5 | 10
  Greece | 8 | 5 | 13
  Thailand | 10 | 9 | 19
  Indonesia | 2 | 0 | 2
  Turkey | 3 | 1 | 4
  Russian Federation | 1 | 1 | 2
  India | 15 | 14 | 29
  Canada | 5 | 3 | 8
  Brazil | 13 | 13 | 26
  Poland | 3 | 5 | 8
  Singapore | 3 | 5 | 8
  South Africa | 3 | 4 | 7
  France | 2 | 0 | 2
  United Kingdom | 0 | 1 | 1
Child-Pugh Class [Number; unit: Participants] — The Child-Pugh classification is used to assess the prognosis of chronic liver disease. The score employs 5 clinical measures of liver disease; each measure is scored 1-3, with 3 indicating most severe derangement. Total possible score is 15. Chronic liver disease is classified into Child-Pugh class A to C, employing the added score from above: 5-6=Class A; 7-9=Class B; 10-15=Class C. As-Randomized population.
  Participants
    Class A | 7 | 10 | 17
    Class B | 63 | 61 | 124
    Class C | 30 | 20 | 50
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] — As-randomized population
  U/L | 99.2 (111.23) | 100.0 (81.68) | 99.6 (98.01)
Child-Pugh Score [Mean (Standard Deviation); unit: units on a scale] — The Child-Pugh classification is used to assess the prognosis of chronic liver disease. The score employs 5 clinical measures of liver disease; each measure is scored 1-3, with 3 indicating most severe derangement. Total possible score is 15. Chronic liver disease is classified into Child-Pugh class A to C, employing the added score from above: 5-6=Class A; 7-9=Class B; 10-15=Class C. As-Randomized population.
  units on a scale | 8.81 (1.98) | 8.35 (1.82) | 8.59 (1.91)
HBV DNA by PCR [Mean (Standard Deviation); unit: log10 copies/mL] — HBV=hepatitis B virus, PCR=polymerase chain reaction. As-Randomized population.
  log10 copies/mL | 7.53 (1.829) | 8.16 (2.179) | 7.83 (2.023)
Mayo End-Stage Liver Disease (MELD) score [Mean (Standard Deviation); unit: units on a scale] — The Model for End-Stage Liver Disease (MELD), is a scoring system for assessing the severity of chronic liver disease. MELD uses the patient's values for serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) to predict survival. In interpreting the MELD Score in hospitalized patients, the 3 month mortality is: 40 or more=100% mortality; 30-39=83% mortality; 20-29=76% mortality; 10-19=27% mortality; <10=4% mortality. As-randomized population.
  units on a scale | 17.07 (5.00) | 15.30 (4.61) | 16.23 (4.89)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hepatitis B Virus (HBV) DNA by Polymerase Chain Reaction (PCR) at Week 24
Description: Mean reduction in serum HBV DNA determined by PCR assay (log10 copies/mL) at Week 24 adjusted for baseline HBV DNA and lamivudine resistance (LVDr) status, based on linear regression analysis.
Time Frame: Baseline, Week 24
Population: Treated Subjects - As-Randomized, modified intention-to-treat (ITT) efficacy data set. Includes on-treatment data (obtained after the start of therapy and no more than 5 days after the last dose of study therapy) collected for treated subjects. Includes those participants with PCR measurements in the Week 24 analysis window.
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 76 | 73
log10 copies/mL | -4.48 (0.200) | -3.40 (0.255)
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Linear regression model adjusted for baseline HBV DNA and LVDr status; Mean Difference (Final Values) = -1.74, 95% CI 2-sided [-2.30 to -1.18]

2. Secondary Outcome: Change From Baseline in HBV DNA by PCR at Week 48
Description: Mean change from baseline in HBV DNA by PCR at Week 48, adjusted for baseline HBV DNA and LVDr Status.
Time Frame: Baseline, Week 48
Population: Treated Subjects - As-Randomized, modified intention-to-treat (ITT) efficacy data set. Includes on-treatment data (obtained after the start of therapy and no more than 5 days after the last dose of study therapy) collected for treated subjects. Includes those participants with PCR measurements in the Week 48 analysis window.
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 69 | 61
log10 copies/mL | -4.66 (0.204) | -3.90 (0.353)
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Test type: Superiority or Other; p < 0.0001, Regression, Linear; adjusted for baseline HBV DNA and LVDr Status; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-1.85 to -0.96]

3. Secondary Outcome: Number of Participants With HBV DNA < 300 Copies/mL by PCR At Week 24
Time Frame: Week 24
Population: Treated Subjects - As-Randomized population, responders only (non-completer=failure).
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
participants | 49 | 15
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Percent Difference = 32.7, 95% CI 2-sided [20.2 to 45.2]

4. Secondary Outcome: Number of Participants With HBV DNA < 300 Copies/mL by PCR At Week 48
Time Frame: Week 48
Population: Treated Subjects - As-Randomized population, responders only (non-completer=failure).
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
Participants | 57 | 18
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean percent treatment difference = 38, 95% CI 2-sided [24.8 to 50.3]

5. Secondary Outcome: Number of Participants Achieving Alanine Transaminase (ALT) Normalization (≤1.0 x Upper Limit of Normal [ULN]) at Weeks 24 and 48
Description: Number of participants in each group who achieved ALT normalization (≤1.0 x upper limit of normal [ULN]) among those with baseline ALT >1.0 x ULN at Weeks 24 and 48
Time Frame: Week 24, Week 48
Population: Treated Subjects - As-Randomized population, responders only (non-completer=failure).Participants in each group who achieved ALT normalization among those with baseline ALT >1.0 x ULN.
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 78 | 71
Participants
  Week 24 | 46 | 28
  Week 48 | 49 | 33
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Week 24 treatment difference; Test type: Superiority or Other; p = 0.0193, Cochran-Mantel-Haenszel; percent treatment difference = 19.2, 95% CI 2-sided [3.7 to 34.6]
Statistical Analysis 2: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Week 48 treatment difference; Test type: Superiority or Other; p = 0.0425, Cochran-Mantel-Haenszel; percent treatment difference = 16.4, 95% CI 2-sided [0.9 to 32.0]

6. Secondary Outcome: Number of Subjects Achieving Composite Endpoint (HBV DNA < 10*4 Copies/mL by PCR Assay and Normal ALT [≤ 1.0 x ULN]) Through Week 48
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 48
Population: Treated Subjects - As-Randomized, modified intention-to-treat (ITT) efficacy data set (includes on-treatment data collected for treated subjects. On-treatment data are those obtained after the start of therapy and no more than 5 days after the last dose of study therapy.) n=number of participants with measurement at baseline and timepoint.
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
Participants
  Baseline | 3 | 1
  Week 4 | 23 | 6
  Week 8 | 34 | 11
  Week 12 | 37 | 16
  Week 24 | 49 | 24
  Week 48 | 57 | 34

7. Secondary Outcome: >=2-Point Reduction From Baseline in Child-Pugh Score Through Week 48
Description: Child-Pugh classification assesses the prognosis of chronic liver disease by 5 clinical measures, scored 1-3 each (most severe derangement=3). Score range: 5 (best prognosis) to 15 (worst prognosis).
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: Treated Subjects-As-Randomized, modified intention-to-treat (ITT) efficacy data set (includes on-treatment data collected for treated subjects. On-treatment data are those obtained after start of therapy and <=5 days after the last dose of study therapy.) Non-completer=Failure. n=number of participants with measurement at baseline and timepoint.
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
Participants
  Baseline | 0 | 0
  Week 4 | 14 | 11
  Week 8 | 23 | 10
  Week 12 | 22 | 11
  Week 24 | 32 | 22
  Week 36 | 35 | 19
  Week 48 | 35 | 25

8. Secondary Outcome: Number of Participants With Improvement or No Worsening in Child-Pugh Score From Baseline to Week 48
Description: Number of participants in each group with improvement or no worsening in Child-Pugh score from baseline to Week 48 as measured by improvement or no worsening in Child-Pugh score. Child-Pugh classification assesses the prognosis of chronic liver disease by 5 clinical measures, scored 1-3 each (most severe derangement=3). Score range: 5 (best prognosis) to 15 (worst prognosis).
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 48
Population: Treated participants (as-randomized). Non-completer=Failure. The modified intention-to-treat (ITT) efficacy data set included on-treatment data collected for treated subjects. On-treatment data are those obtained after the start of therapy and no more than 5 days after the last dose of study therapy.
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
Participants
  Baseline | 0 | 0
  Week 4 | 66 | 67
  Week 8 | 67 | 62
  Week 12 | 68 | 62
  Week 24 | 66 | 65
  Week 48 | 61 | 61

9. Secondary Outcome: Change From Baseline in Child-Pugh Score Through Week 48
Description: Mean change from baseline in Child-Pugh score through week 48. Child-Pugh classification assesses the prognosis of chronic liver disease by 5 clinical measures, scored 1-3 each (most severe derangement=3). Score range: 5 (best prognosis) to 15 (worst prognosis).
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: as for outcome 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
units on a scale
  Baseline Value (n=100, n=91) | 8.8 (0.20) | 8.4 (0.19)
  Change at Week 4 (n=90; n=85) | -0.4 (0.14) | -0.3 (0.14)
  Change at Week 8 (n=90; n=79) | -0.4 (0.18) | -0.3 (0.17)
  Change at Week 12 (n=87; n=80) | -0.6 (0.18) | -0.3 (0.15)
  Change at Week 24 (n=80; n=77) | -1.2 (0.20) | -0.7 (0.18)
  Change at Week 36 (n=75; n=70) | -1.6 (0.25) | -0.9 (0.18)
  Change at Week 48 (n=72; n=64) | -1.7 (0.26) | -1.3 (0.19)

10. Secondary Outcome: Number of Participants With Improvement in Child-Pugh Class at Week 24 and Week 48
Description: Number of Participants in each group with improvement in Child-Pugh score from baseline to Week 48 as measured by improvement in Child-Pugh class. Improvement in Child-Pugh Class is defined as change from B to A or C to A. Evaluable subjects are subjects with Child-Pugh Class B or C at Baseline. Child-Pugh classification assesses the prognosis of chronic liver disease by 5 clinical measures, scored 1-3 each (most severe derangement=3). Score range: 5 (best prognosis) to 15 (worst prognosis). Child-Pugh class A to C employs the added score from above: 5-6=Class A; 7-9=Class B; 10-15=Class C.
Time Frame: Week 24, Week 48
Population: Treated participants (as-randomized). The modified intention-to-treat (ITT) efficacy data set included on-treatment data collected for treated subjects. On-treatment data are those obtained after the start of therapy and no more than 5 days after the last dose of study therapy.
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 93 | 81
Participants
  Week 24 | 25 | 22
  Week 48 | 35 | 29

11. Secondary Outcome: Mean Change From Baseline in Model for End-Stage Liver Disease (MELD) Scores From Baseline Through Week 48
Description: Adjusted mean change from baseline in MELD score through Week 48 (adjusted for baseline value). The Model for End-Stage Liver Disease (MELD), is a scoring system for assessing the severity of chronic liver disease. MELD uses the patient's values for serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) to predict survival. In interpreting the MELD Score in hospitalized patients, the 3 month mortality is: 40 or more=100% mortality; 30-39=83% mortality; 20-29=76% mortality; 10-19=27% mortality; <10=4% mortality.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: Treated participants - as-randomized populations; n=number of participants with assessment at baseline and timepoint. The modified intention-to-treat (ITT) efficacy data set included on-treatment data collected for treated subjects. On-treatment data are obtained after the start of therapy and <=5 days after the last dose of study therapy.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
units on a scale
  Baseline Value (n=100; n=91) | 17.1 (0.50) | 15.3 (0.48)
  Week 4 (n=97; n=87) | -0.1 (0.38) | 0.1 (0.25)
  Week 8 (n=90; n=79) | -0.8 (0.35) | -0.4 (0.34)
  Week 12 (n=88; n=80) | -1.2 (0.41) | -0.9 (0.32)
  Week 24 (n=80; n=77) | -2.0 (0.45) | -0.9 (0.46)
  Week 36 (n=75; n=70) | -2.3 (0.57) | -1.2 (0.48)
  Week 48 (n=72; n=62) | -2.6 (0.62) | -1.7 (0.50)
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Covariate adjusted model for MELD score at Week 24; Test type: Superiority or Other; p = 0.51, Regression, Linear; Model estimate incorporates prognostic factors measured at baseline. Adjusted for baseline; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-1.63 to 0.82]
Statistical Analysis 2: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Covariate adjusted model for MELD score at Week 48; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Model estimate incorporates prognostic factors measured at baseline. Adjusted for baseline; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-1.08 to 1.88]

12. Secondary Outcome: Improvement or No Worsening in MELD Score Through Week 48
Description: Participants with improvement or no worsening (any decrease or no change from baseline in score) in MELD score through Week 48. The Model for End-Stage Liver Disease (MELD), is a scoring system for assessing the severity of chronic liver disease. MELD uses the patient's values for serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) to predict survival. In interpreting the MELD Score in hospitalized patients, the 3 month mortality is: 40 or more=100% mortality; 30-39=83% mortality; 20-29=76% mortality; 10-19=27% mortality; <10=4% mortality.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 48
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
Participants
  Baseline | 0 | 0
  Week 4 | 58 | 51
  Week 8 | 63 | 52
  Week 12 | 67 | 60
  Week 24 | 62 | 51
  Week 48 | 53 | 47

13. Secondary Outcome: Mean Changes From Baseline in Quality of Life as Measured by the Short Form 36 (SF-36)
Description: Scoring for the SF-36 will be done using the algorithm developed by the Research ANd Development(RAND) Corporation (a scale of 0-100). Higher scores represent better quality of life. Coding for items with 2-category responses=0 and 100; 3-category=0/50/100; 5-category=0/25/50/75/100; 6-category=0/20/40/60/80/100. Scores of items in the same scale are combined to create the 8 scale scores (physical functioning, role-physical, bodily-pain, general health, vitality, social functioning, role-emotional, mental health). Physical and mental health composite scores will be computed for the group.
Time Frame: Baseline, Week 24, Week 48
Population: This endpoint was not analyzed due to lack of complete data at 48 Weeks, but will be assessed at future time points.
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Mean Changes From Baseline in Quality of Life, as Measured by EuroQol-5D (EQ-5D) at Weeks 24 and 48
Description: The EQ-5D has 5 attributes (mobility, self-care, usual activity, pain/discomfort, and anxiety/depression), each with 3 levels (no problem, some problems, and major problems). This algorithm gives valuation (weights) to each of the 15 responses on the form. Each valuation is a negative number, subtracted from the maximum score of 1 (perfect well being). The overall health index score ranges from 0 (dead) to 1 (perfect health) value scale, and the visual analog scale ranges from 0 to 100. Item weights will be obtained from the EuroQol group.
Time Frame: Baseline, Week 24, Week 48
Population: This endpoint was not analyzed due to lack of complete data at 48 Weeks, but will be assessed at future time points.
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change From Baseline in Albumin Through Week 48
Description: Mean albumin levels, and mean change from baseline in albumin, a measure of synthetic liver function. Normal range for albumin = 3.5 - 5.3 g/dL.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: Treated participants - as randomized; n=number of participants with value at baseline and given timepoint.
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
g/dL
  Baseline Value (n=100; n=91) | 3.00 (0.55) | 3.10 (0.067)
  Change at Week 4 (n=98; n=88) | -0.04 (0.032) | -0.01 (0.033)
  Change at Week 8 (n=92; n=82) | 0.01 (0.034) | -0.03 (0.037)
  Change at Week 12 (n=88; n=80) | 0.05 (0.039) | 0.03 (0.037)
  Change at Week 24 (n=81; n=77) | 0.26 (0.056) | 0.20 (0.048)
  Change at Week 36 (n=76; n=70) | 0.36 (0.062) | 0.25 (0.052)
  Change at Week 48 (n=72; n=63) | 0.49 (0.061) | 0.34 (0.057)

16. Secondary Outcome: Mean Change From Baseline in Prothrombin Time Through Week 48
Description: Mean prothrombin time, and mean change from baseline in prothrombin time, a measure of synthetic liver function. Prothrombin time is the time it takes (in seconds) for a sample of blood to clot. Normal range for prothrombin time (PT) = 10-13 seconds.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: Treated, as-randomized. Subjects with normal values at baseline were excluded from the analysis. n=number of participants with value at baseline and given timepoint.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
seconds
  Baseline Value (n=100; n=91) | 16.28 (0.234) | 15.35 (0.196)
  Change at Week 4 (n=98; n=87) | -0.08 (0.156) | 0.03 (0.114)
  Change at Week 8 (n=91; n=79) | -0.10 (0.158) | 0.06 (0.161)
  Change at Week 12 (n=88; n=80) | -0.29 (0.153) | -0.05 (0.162)
  Change at Week 24 (n=80; n=77) | -0.75 (0.216) | -0.18 (0.205)
  Change at Week 48 (n=72; n=63) | -0.99 (0.288) | -0.52 (0.197)

17. Secondary Outcome: Mean Change From Baseline in Total Bilirubin Through Week 48
Description: Mean total bilirubin levels, and mean change from baseline in total bilirubin, a measure of liver secretory function.Normal range for total bilirubin = 0.2 - 1.2 mg/dL.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: as for outcome 16
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 100 | 91
mg/dL
  Baseline Value (n=100; n=91) | 2.80 (0.207) | 2.50 (0.214)
  Change at Week 4 (n=98; n=88) | -0.06 (0.154) | 0.21 (0.172)
  Change at Week 8 (n=92; n=82) | 0.11 (0.376) | -0.17 (0.094)
  Change at Week 12 (n=88;l n=80) | -0.20 (0.193) | -0.28 (0.109)
  Change at Week 24 (n=81; n=77) | -0.41 (0.154) | -0.14 (0.227)
  Change at Week 36 (n=76; n=70) | -0.36 (0.329) | -0.09 (0.298)
  Change at Week 48 (n=72; n=63) | -0.61 (0.233) | -0.10 (0.450)

18. Secondary Outcome: Change From Baseline in Platelet Count Through Week 48
Description: Mean baseline platelet count and mean change from baseline in platelet count at specific timepoints. Platelets are the smallest particles found in the blood, which play a major role in forming blood clots. Normal range for platelets = 140 - 450 X 10*9 c/L.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: as for outcome 16
Measure: Mean (Standard Error); unit: 10*9 c/L
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 97 | 91
10*9 c/L
  Baseline Value (n=97; n=91) | 87.32 (4.771) | 93.31 (4.947)
  Change at Week 4 (n=90; n=85) | -0.93 (2.064) | -2.14 (2.553)
  Change at Week 8 (n=82; n=76) | 3.55 (3.063) | 3.88 (2.923)
  Change at Week 12 (n=85; n=79) | 4.36 (2.837) | -0.81 (2.814)
  Change at Week 24 (n=77; n=76) | 2.47 (2.556) | -2.89 (3.205)
  Change at Week 36 (n=72; n=69) | 6.56 (3.534) | 1.32 (3.188)
  Change at Week 48 (n=68; n=63) | 10.19 (4.956) | 3.05 (3.570)

19. Secondary Outcome: Participants Achieving Albumin Normalization Through Week 48
Description: Number of participants who achieved normalization of albumin (>= 1 x lower limit of normal [LLN]), a measure of liver function, at specific timepoints.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: Treated subjects (as randomized). Excludes subjects with normal albumin at Baseline. Non-completer = failure.
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 82 | 69
participants
  Baseline | 0 | 0
  Week 4 | 2 | 7
  Week 8 | 9 | 6
  Week 12 | 6 | 11
  Week 24 | 20 | 14
  Week 36 | 29 | 14
  Week 48 | 32 | 20
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Difference estimate ETV - ADV at Week 48; Test type: Superiority or Other; Difference Estimate = 10.4, 95% CI 2-sided [-4.5 to 25.2]

20. Secondary Outcome: Participants Achieving Prothrombin Time Normalization Through Week 48
Description: Number of participants who achieved normalization of prothrombin time (<= 1 x ULN), a measure of liver function, at specific timepoints.
Time Frame: Baseline, Week4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: Treated subjects - as-randomized. Excludes participants with normal prothrombin time at baseline. Non-completer = failure.
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 95 | 82
participants
  Baseline | 0 | 0
  Week 4 | 3 | 4
  Week 8 | 5 | 4
  Week 12 | 4 | 3
  Week 24 | 9 | 6
  Week 36 | 10 | 5
  Week 48 | 8 | 7
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Difference Estimate at Week 48; Test type: Superiority or Other; Difference Estimate = -0.4, 95% CI 2-sided [-8.7 to 8.0]

21. Secondary Outcome: Participants Achieving Total Bilirubin Normalization Through Week 48
Description: Number of participants who achieved normalization of total bilirubin (<= 1 x ULN), a measure of liver function, at specific timepoints.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 75 | 65
participants
  Baseline | 0 | 0
  Week 4 | 4 | 9
  Week 8 | 10 | 9
  Week 12 | 8 | 9
  Week 24 | 12 | 10
  Week 36 | 9 | 17
  Week 48 | 15 | 18
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Difference Estimate at Week 48; Test type: Superiority or Other; Difference Estimate = -7.2, 95% CI 2-sided [-21.3 to 6.9]

22. Secondary Outcome: Participants Achieving Platelet Count Normalization Through Week 48
Description: Number of participants who achieved normalization of platelet count (>= 1 x lower limit of normal [LLN]), a measure of liver function, at specific timepoints.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 85 | 76
participants
  Baseline | 0 | 0
  Week 4 | 3 | 4
  Week 8 | 3 | 5
  Week 12 | 7 | 3
  Week 24 | 2 | 2
  Week 36 | 5 | 2
  Week 48 | 6 | 1
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; Difference Estimate at Week 48; Test type: Superiority or Other; Difference Estimate = 5.7, 95% CI 2-sided [-0.3 to 11.7]

23. Secondary Outcome: Number of Hepatocellular Carcinoma (HCC) Events at Different Time Points Through Week 48
Description: HCC-free survival was analyzed using life tables. Measured values show the number of HCC events among treated participants at given time points.
Time Frame: Week 48
Population: Treated, through Week 48 - (analyzed as-treated). (Week 48 on-treatment safety data contain all on-treatment data up to study Day 336, if the subject is still on treatment. If the subject discontinued before study Day 336, then all data up to 5 days after the discontinuation date were included.) n=number of participants at risk at each timepoint.
Measure: Number; unit: HCC events
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 102 | 89
HCC events
  Weeks 0-4 (n=102; n=89) | 2 | 3
  Weeks 4-8 (n=99; n=86) | 5 | 5
  Weeks 8-12 (n=96; n=83) | 10 | 6
  Weeks 12-16 (n=90; n=80) | 11 | 9
  Weeks 16-20 (n=87; n=77) | 11 | 11
  Weeks 20-24 (n=86; n=75) | 16 | 14
  Weeks 24-28 (n=81; n=71) | 17 | 15
  Weeks 28-32 (n=78; n=70) | 17 | 17
  Weeks 32-36 (n=77; n=66) | 17 | 18
  Weeks 36-40 (n=77; n=64) | 19 | 20
  Weeks 40-44 (n=73; n=62) | 21 | 20
  Weeks 44-48 (n=71; n=62) | 24 | 22
Statistical Analysis 1: Comparison: Entecavir (ETV) 1.0 mg vs Adefovir (ADV) 10 mg; treatment comparison of HCC-free survival at Week 48; Test type: Superiority or Other; p = 0.20, Regression, Cox; Cox proportional hazard model, adjusted for age <=45 versus age >45 years, gender, and race (white versus non-white); Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.46 to 1.18]

24. Secondary Outcome: Cumulative Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, HCC, Discontinuations Due to AEs, and Confirmed Creatinine Increase >=0.5 mg/dL
Description: AE=any new untoward medical occurrence/worsening of a pre-existing medical condition regardless of causal relationship. SAE=any untoward medical occurrence at any dose that: results in death; is life-threatening; requires/prolongs inpatient hospitalization; results in persistent/significant disability; is cancer; is congenital anomaly/birth defect; results in drug dependency/abuse; is an important medical event. Grades:1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death. Confirmed increase in serum creatinine=values ≥0.5 mg/dL compared with baseline on 2 sequential measures.
Time Frame: on-treatment events obtained after the start of therapy and no more than 5 days after the last dose of study therapy.
Population: As-treated population (all randomized subjects treated with at least 1 dose of study therapy, ETV or ADV, based on actual treatment received). Note that 5 additional enrolled participants died prior to initiation of treatment and are not included in this table.
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 102 | 89
participants
  Any AE | 91 | 86
  Grade 3/4 AEs | 55 | 42
  SAEs | 70 | 59
  Deaths | 23 | 29
  HCC | 12 | 18
  Discontinuations due to AEs | 7 | 5
  Confirmed creatinine increase >= 0.5 mg/dL | 17 | 21

25. Secondary Outcome: Number of Participants With Treatment-Emergent Grade 3/4 Laboratory Abnormalities - Week 48 and Cumulative Data
Description: Grade 3/4 laboratory abnormalities (hematology, electrolyte, lipase, liver function, metabolic, renal function, urinalysis). The Week 48 data set was used to evaluate the Week-48 on-treatment safety. The cumulative data set was used to evaluate the safety while on treatment. Common Terminology Criteria for Adverse Events v3.0 (CTCAE) Grades:1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death.
Time Frame: Week 48=all on-treatment laboratory measurements up to Week 48. Cumulative data = on-treatment laboratory measurements obtained after the start of therapy and no more than 5 days after the last dose of study therapy.
Population: As-treated population (all randomized subjects treated with at least 1 dose of study therapy, ETV or ADV, based on actual treatment received).
Measure: Number; unit: participants
Arm/Group | Week 48 - Entecavir (ETV) 1.0 mg | Week 48 - Adefovir (ADV) 10 mg | Cumulative - Entecavir (ETV) 1.0 mg | Cumulative - Adefovir (ADV) 10 mg
Number analyzed (Participants) | 102 | 89 | 102 | 89
participants
  Hemoglobin | 8 | 8 | 11 | 10
  International Normalized Ratio | 30 | 22 | 40 | 32
  Platelet Count | 20 | 21 | 25 | 24
  Prothrombin Time | 20 | 7 | 25 | 11
  Bicarbonate, Low | 3 | 4 | 4 | 4
  Chloride, Serum, Low | 2 | 2 | 2 | 2
  Bicarbonate/Carbon Dioxide, Low | 3 | 4 | 4 | 4
  Potassium, Serum, High | 1 | 0 | 1 | 0
  Sodium, Serum | 6 | 3 | 6 | 5
  Sodium, Serum, Low | 6 | 3 | 6 | 5
  Lipase, Total (colorimetric assay) | 17 | 18 | 23 | 25
  Alanine Aminotransferase (ALT) | 3 | 1 | 5 | 4
  Albumin | 9 | 3 | 9 | 3
  Alkaline Phosphatase (ALP) | 0 | 1 | 1 | 1
  Aspartate Aminotransferase (AST) | 7 | 3 | 9 | 7
  Bilirubin, Total | 19 | 18 | 24 | 25
  G-Glutamyl Transferase (GGT) | 1 | 6 | 9 | 10
  Glucose, Fasting Serum, High | 0 | 0 | 1 | 0
  Creatinine | 1 | 0 | 2 | 0
  Phosphorus, inorganic | 0 | 4 | 0 | 6
  Blood, urine | 13 | 13 | 18 | 22
  Glucose, urine | 11 | 11 | 17 | 13
  Protein, urine | 1 | 2 | 2 | 4
  Neutrophils (relative) | 0 | 1 | 0 | 1
  Neutrophils + Bands (relative) | 2 | 4 | 4 | 8
  Neutrophils (absolute) | 2 | 3 | 5 | 7

26. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Flares - On Treatment
Description: ALT flare=ALT > 2 x baseline and > 10 x upper limit of normal (ULN) by clinical laboratory evaluation. Table includes number of participants with selected clinical events and/or laboratory abnormalities during ALT flares. Selected clinical events during ALT flares=ascites, hepatic encephalopathy, jaundice, bacterial peritonitis. Selected Laboratory abnormalities during ALT flares=international normalized ratio > 1.5 or prothrombin time >= 1.2 x ULN and total bilirubin >2.5 mg/dL and > 1 mg/dL increase from baseline.
Time Frame: On-treatment=up to Week 48 (Day 336); if discontinued early, all data up to 5 days after discontinuation date.
Population: Treated participants - as treated. The on-treatment safety data set contains data from all randomized subjects treated with at least 1 dose of study therapy, ETV or ADV. Treatment group for safety data set is based on actual treatment received.
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 102 | 89
participants
  ALT flares | 2 | 1
  ALT flares, no clinical events/lab abnormalities | 1 | 0
  ALT flares, with clinical events/lab abnormalities | 1 | 1

27. Secondary Outcome: Number of Participants With Malignant Neoplasms - On Treatment or During 24-Week Follow-up Period
Description: Data includes type of malignant neoplasm.
Time Frame: On-treatment=up to Week 48 (Day 336); if discontinued early, all data up to 5 days after discontinuation date. 24-week follow-up=limited to end-of-dosing values and those from 6 days after last dose of study therapy to end of follow-up.
Population: The on-treatment safety data set contains data from all randomized subjects treated with at least 1 dose of study therapy, ETV or ADV. Treatment group for safety data set is based on actual treatment received.
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 102 | 89
participants
  Any Adverse Events | 14 | 18
  Hepatic Neoplasm, Malignant | 12 | 18
  Basal Cell Carcinoma | 1 | 0
  Lymph Node Cancer, Metastatic | 1 | 0
  Hepatic Mass | 1 | 0

28. Secondary Outcome: Number of Participants Undergoing Liver Transplant - On-Treatment or 24-Week Follow-Up
Time Frame: as for outcome 27
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | Entecavir (ETV) 1.0 mg | Adefovir (ADV) 10 mg
Number analyzed (Participants) | 102 | 89
participants
  Liver Transplant: Yes | 11 | 3
  Liver Transplant: No | 91 | 86

ADVERSE EVENTS:
Arm/Group | ADEFOVIR | ENTECAVIR
Serious Adverse Events (participants affected / at risk) | 59/89 | 70/102
Other Adverse Events (participants affected / at risk) | 76/89 | 77/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADEFOVIR (N=89) | ENTECAVIR (N=102)
CATARACT (Eye disorders) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
BLOOD ALBUMIN DECREASED (Investigations) | 2 | 2
HEPATIC ENZYME INCREASED (Investigations) | 1 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 6 | 8
PROTHROMBIN TIME ABNORMAL (Investigations) | 2 | 3
BLOOD CREATININE INCREASED (Investigations) | 1 | 0
PROTHROMBIN TIME PROLONGED (Investigations) | 13 | 14
BLOOD BICARBONATE DECREASED (Investigations) | 0 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
INTERNATIONAL NORMALISED RATIO ABNORMAL (Investigations) | 1 | 2
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 5 | 5
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0
BLEEDING VARICOSE VEIN (Vascular disorders) | 1 | 1
CARDIOVASCULAR INSUFFICIENCY (Vascular disorders) | 0 | 1
ALCOHOL USE (Social circumstances) | 1 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 2 | 0
HEPATIC MASS (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 2
LIVER DISORDER (Hepatobiliary disorders) | 1 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 2 | 10
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 3 | 3
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 2 | 0
PORTAL HYPERTENSION (Hepatobiliary disorders) | 1 | 0
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 3 | 3
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
HEPATITIS CHOLESTATIC (Hepatobiliary disorders) | 0 | 1
CHRONIC HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 2
HEPATIC ARTERY THROMBOSIS (Hepatobiliary disorders) | 1 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 2 | 2
TRANSPLANT REJECTION (Immune system disorders) | 0 | 1
LIVER TRANSPLANT REJECTION (Immune system disorders) | 0 | 1
COMA HEPATIC (Nervous system disorders) | 0 | 1
HYDROCEPHALUS (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 3 | 2
SENSORY DISTURBANCE (Nervous system disorders) | 0 | 1
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 9 | 10
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 0
ASCITES (Gastrointestinal disorders) | 4 | 4
MELAENA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 2
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 2
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 2
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
LEUKOPLAKIA ORAL (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRITIS ALCOHOLIC (Gastrointestinal disorders) | 1 | 0
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 0 | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRIC VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 4 | 0
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 2 | 4
PORTAL HYPERTENSIVE GASTROPATHY (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 4
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 1
OTOTOXICITY (Ear and labyrinth disorders) | 1 | 0
SEPSIS (Infections and infestations) | 3 | 5
PNEUMONIA (Infections and infestations) | 2 | 3
UROSEPSIS (Infections and infestations) | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 3
BACTERAEMIA (Infections and infestations) | 1 | 0
HEPATITIS B (Infections and infestations) | 1 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 1 | 4
GASTROENTERITIS (Infections and infestations) | 0 | 2
SCROTAL INFECTION (Infections and infestations) | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1
TESTICULAR ABSCESS (Infections and infestations) | 0 | 1
PERINEPHRIC ABSCESS (Infections and infestations) | 0 | 1
NECROTISING FASCIITIS (Infections and infestations) | 0 | 1
PERITONITIS BACTERIAL (Infections and infestations) | 6 | 6
PULMONARY TUBERCULOSIS (Infections and infestations) | 2 | 0
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 | 1
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 | 0
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0
GASTRIC ULCER HELICOBACTER (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
BETA HAEMOLYTIC STREPTOCOCCAL INFECTION (Infections and infestations) | 0 | 1
ANURIA (Renal and urinary disorders) | 1 | 0
OLIGURIA (Renal and urinary disorders) | 0 | 1
CALCULUS BLADDER (Renal and urinary disorders) | 1 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 1
CHOLECYSTECTOMY (Surgical and medical procedures) | 1 | 0
LIVER TRANSPLANT (Surgical and medical procedures) | 0 | 7
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 3
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 1
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 1
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1
EXOMPHALOS (Congenital, familial and genetic disorders) | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 1
TESTICULAR INJURY (Injury, poisoning and procedural complications) | 0 | 1
FOREIGN BODY TRAUMA (Injury, poisoning and procedural complications) | 1 | 0
FASCIITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 2
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HEPATIC HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DEATH (General disorders) | 0 | 2
PYREXIA (General disorders) | 3 | 2
ASTHENIA (General disorders) | 0 | 1
CHEST PAIN (General disorders) | 1 | 0
SUDDEN DEATH (General disorders) | 0 | 1
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 | 1
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 12
LYMPH NODE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEPATIC NEOPLASM MALIGNANT RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADEFOVIR (N=89) | ENTECAVIR (N=102)
HYPERTENSION (Vascular disorders) | 4 | 10
INSOMNIA (Psychiatric disorders) | 8 | 9
HEADACHE (Nervous system disorders) | 18 | 7
DIZZINESS (Nervous system disorders) | 9 | 9
ENCEPHALOPATHY (Nervous system disorders) | 1 | 7
NAUSEA (Gastrointestinal disorders) | 4 | 11
ASCITES (Gastrointestinal disorders) | 14 | 14
VOMITING (Gastrointestinal disorders) | 8 | 12
DIARRHOEA (Gastrointestinal disorders) | 18 | 15
DYSPEPSIA (Gastrointestinal disorders) | 6 | 10
TOOTHACHE (Gastrointestinal disorders) | 6 | 3
CONSTIPATION (Gastrointestinal disorders) | 6 | 9
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 | 14
DUODENAL ULCER (Gastrointestinal disorders) | 7 | 3
GINGIVAL BLEEDING (Gastrointestinal disorders) | 2 | 6
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 6 | 4
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 7 | 7
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 9 | 12
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 | 3
INFLUENZA (Infections and infestations) | 5 | 8
PNEUMONIA (Infections and infestations) | 2 | 7
CELLULITIS (Infections and infestations) | 5 | 2
NASOPHARYNGITIS (Infections and infestations) | 9 | 8
URINARY TRACT INFECTION (Infections and infestations) | 6 | 7
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 14 | 19
HAEMATURIA (Renal and urinary disorders) | 7 | 1
ANOREXIA (Metabolism and nutrition disorders) | 5 | 4
DIABETES MELLITUS (Metabolism and nutrition disorders) | 5 | 5
ANAEMIA (Blood and lymphatic system disorders) | 5 | 6
PRURITUS (Skin and subcutaneous tissue disorders) | 5 | 7
GYNAECOMASTIA (Reproductive system and breast disorders) | 2 | 10
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 | 8
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 4
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 15 | 17
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 5
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5 | 9
FATIGUE (General disorders) | 13 | 13
PYREXIA (General disorders) | 16 | 20
ASTHENIA (General disorders) | 7 | 7
CHEST PAIN (General disorders) | 5 | 5
OEDEMA PERIPHERAL (General disorders) | 21 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.